CLINICAL TRIAL: NCT03805113
Title: Efficacy of Magnetotherapy in Hand Erosive Osteoarthritis. A Randomized Clinical Trial.
Brief Title: Efficacy of Magnetotherapy in Hand Erosive Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Principal Investigator, Anna Boada-Pladellorens, MD, Hospital Mutua de Terrassa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02/16
Record Dates: First submitted 2019-01-10; First posted 2019-01-15 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Musculoskeletal Disease; Musculoskeletal Pain; Physical Therapy
Keywords: Erosive arthritis; Hands arthritis; Magnetotherapy
MeSH Terms: conditions — Musculoskeletal Diseases; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Treatment with magnetotherapy device 15 20-minute-sesions every consecutive working day.
  Interventions: Device: Magnetotherapy device
- Control group placebo (Placebo Comparator): Treatment with misconnected magnetotherapy device 15 20-minute-sesions every consecutive working day.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Magnetotherapy device — Use of magnetotherapy device 15 consecutive working days in elegible patients with erosive hand osteoarthritis.
  Arms: Intervention group
Device: Placebo — Use of unplugged magnetotherapy device 15 consecutive working days in elegible patients with erosive hand osteoarthritis.
  Arms: Control group placebo

SUMMARY:
Erosive arthritis (EA) is an unusual pathology. There is no definitive treatment and the conventional one has little efficacy. Despite using magnetotherapy (MGT) as a treatment, there is no evidence supporting its use.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the efficacy of MGT in patients suffering from hand EA, compared to placebo, in terms of pain (assessed by Visual Analog Scale (VAS)) and functionality (assessed by The Disabilities of the Arm, Shoulder and Hand (DASH) score) during the treatment and after a 3-months period. Secondarily, rigidity (Modified Kapandji Index), grip strength (JAMAR dynamometry) and quality of life (SF-36 questionnaire) were assessed. Treatment safety will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes older than 18 years with symptomatic hand erosive osteoarthritis for more than 6 months.
* Patients receiving treatment or not for their hand pathology.
* Patients suffering from hand chronic pain due to their pathology and scoring VAS equal or greater than 4/10.
* Patients who voluntarily signed the informed consent and agree to participate in the study.

Exclusion Criteria:

* Pregnancy
* Patients with pacemaker or similar devices
* Pacients with cognitive dysfunction.
* Patients with psychiatric pathologies unable to comply with the treatment and follow-up
* Patients with active oncological and / or infectious pathology
* Patients with previous magnetotherapy or paraffin treatment in the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-01-02 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from baseline pain at the end of the intervention and 3 months after the end of intervention.
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which measures subjective characteristics or attitudes that cannot be directly measured, like pain. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points: one meaning no pain and the opposite one meaning the worst pain.

SECONDARY OUTCOMES:
The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | Before starting the intervention, at the end of the intervention and 3 months after the end of intervention.
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.
Modified Kapandji Index | Before starting the intervention, at the end of the intervention and 3 months after the end of intervention.
  Modified Kapandji Index is a rate of hand mobility assessment. The final result is obtained by adding the results of the 3 tests: test opposition of the thumb (It consists of touching the 4 fingers with the thumb pulp. It scores from 0 to 10); fingers flexion test (It consists of following the thumb with each of the fingers, scoring from 0 (impossible to achieve) to 20 (completely achieved)); fingers extension test (It consists of stretching the hand on a table and get the maximum contact with the surface of the table, scoring from 0 (impossible to achieve) to 20 (completely achieved)).
JAMAR dynamometry | Before starting the intervention, at the end of the intervention and 3 months after the end of intervention.
  JAMAR dynamometry is a valid and reliable instrument to measure the muscular strength of the hands. It is needed to be well performed. The patient is placed in a sitting position with the elbows flexed to 90 degrees without supporting them and the JAMAR is approached to him to be able to make 3 strength determinations with each hand. The final value is extracted from the average of the 3 values of each hand.
SF-36 questionnaire | Before starting the intervention, at the end of the intervention and 3 months after the end of intervention.
  SF-36 is a self-administered questionnaire that can be answered in approximately 10 minute. It quantifies thepatients health status using 8 scales that measure three aspects: functional status, well-being and overall health assessment. 8 numbers between 0 and 100 are obtained. The higher score, the better health status is.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Boada-Pladellorens, MD, Principal Investigator — Hospital Nostra Senyora de Meritxell

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kwok WY, Kloppenburg M, Rosendaal FR, van Meurs JB, Hofman A, Bierma-Zeinstra SM. Erosive hand osteoarthritis: its prevalence and clinical impact in the general population and symptomatic hand osteoarthritis. Ann Rheum Dis. 2011 Jul;70(7):1238-42. doi: 10.1136/ard.2010.143016. Epub 2011 Apr 6. PMID 21474485
- [Background] Gazeley DJ, Yeturi S, Patel PJ, Rosenthal AK. Erosive osteoarthritis: A systematic analysis of definitions used in the literature. Semin Arthritis Rheum. 2017 Feb;46(4):395-403. doi: 10.1016/j.semarthrit.2016.08.013. Epub 2016 Aug 24. PMID 27692966
- [Background] Haugen IK, Mathiessen A, Slatkowsky-Christensen B, Magnusson K, Boyesen P, Sesseng S, van der Heijde D, Kvien TK, Hammer HB. Synovitis and radiographic progression in non-erosive and erosive hand osteoarthritis: is erosive hand osteoarthritis a separate inflammatory phenotype? Osteoarthritis Cartilage. 2016 Apr;24(4):647-54. doi: 10.1016/j.joca.2015.11.014. Epub 2015 Nov 24. PMID 26620088
- [Background] Zhang W, Doherty M, Leeb BF, Alekseeva L, Arden NK, Bijlsma JW, Dincer F, Dziedzic K, Hauselmann HJ, Kaklamanis P, Kloppenburg M, Lohmander LS, Maheu E, Martin-Mola E, Pavelka K, Punzi L, Reiter S, Smolen J, Verbruggen G, Watt I, Zimmermann-Gorska I; ESCISIT. EULAR evidence-based recommendations for the diagnosis of hand osteoarthritis: report of a task force of ESCISIT. Ann Rheum Dis. 2009 Jan;68(1):8-17. doi: 10.1136/ard.2007.084772. Epub 2008 Feb 4. PMID 18250111
- [Background] Kanat E, Alp A, Yurtkuran M. Magnetotherapy in hand osteoarthritis: a pilot trial. Complement Ther Med. 2013 Dec;21(6):603-8. doi: 10.1016/j.ctim.2013.08.004. Epub 2013 Sep 8. PMID 24280467
- [Background] Anandarajah A. Erosive osteoarthritis. Discov Med. 2010 May;9(48):468-77. PMID 20515616
- [Background] Gummesson C, Atroshi I, Ekdahl C. The disabilities of the arm, shoulder and hand (DASH) outcome questionnaire: longitudinal construct validity and measuring self-rated health change after surgery. BMC Musculoskelet Disord. 2003 Jun 16;4:11. doi: 10.1186/1471-2474-4-11. Epub 2003 Jun 16. PMID 12809562
- [Background] Spadoni GF, Stratford PW, Solomon PE, Wishart LR. The evaluation of change in pain intensity: a comparison of the P4 and single-item numeric pain rating scales. J Orthop Sports Phys Ther. 2004 Apr;34(4):187-93. doi: 10.2519/jospt.2004.34.4.187. PMID 15128188
- [Background] Garratt AM, Ruta DA, Abdalla MI, Buckingham JK, Russell IT. The SF36 health survey questionnaire: an outcome measure suitable for routine use within the NHS? BMJ. 1993 May 29;306(6890):1440-4. doi: 10.1136/bmj.306.6890.1440. PMID 8518640
- [Background] Lefevre-Colau MM, Poiraudeau S, Oberlin C, Demaille S, Fermanian J, Rannou F, Revel M. Reliability, validity, and responsiveness of the modified Kapandji index for assessment of functional mobility of the rheumatoid hand. Arch Phys Med Rehabil. 2003 Jul;84(7):1032-8. doi: 10.1016/s0003-9993(03)00128-x. PMID 12881830
- [Background] Stark T, Walker B, Phillips JK, Fejer R, Beck R. Hand-held dynamometry correlation with the gold standard isokinetic dynamometry: a systematic review. PM R. 2011 May;3(5):472-9. doi: 10.1016/j.pmrj.2010.10.025. PMID 21570036